CLINICAL TRIAL: NCT01692496
Title: Phase II Clinical Trial of Pazopanib to Evaluate the Activity and Tolerability in Patients With Advanced and/or Metastatic Liposarcoma Who Have Relapsed Following Standard Therapies or for Whom no Standard Therapy Exists
Brief Title: Activity and Tolerability of Pazopanib in Advanced and/or Metastatic Liposarcoma. A Phase II Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-30; 2012-002745-38 (EudraCT Number)
Record Dates: First submitted 2012-09-14; First posted 2012-09-25 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Advanced and / or Metastatic Liposarcoma
Keywords: Advanced; Metastatic; Liposarcoma; Pazopanib
MeSH Terms: conditions — Liposarcoma; Neoplasm Metastasis | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental): Patients will receive oral pazopanib, 800mg once daily and treatment will continue until disease progression, development of unacceptable toxicity, noncompliance, withdrawal of consent by the patient or investigator decision.
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Patients will receive oral pazopanib, 800mg once daily and treatment will continue until disease progression, development of unacceptable toxicity, noncompliance, withdrawal of consent by the patient or investigator decision.

SUMMARY:
Soft tissue and bone sarcomas are rare malignant tumors, which encompasses a large family of more than 50 histologically distinct tumor subtypes, all of which share a putative mesenchymal origin. In the case of soft tissue sarcomas (STS) surgical excision is the mainstay of treatment, but despite curative surgery, around half of patients develop distant metastases and die from disease. Few therapeutic approaches are currently available to patients with unresectable, locally advanced, or metastatic STS and only anthracyclines, ifosfamide and trabectedin have shown activity, with response rates of 20-40% in previously untreated patients. Recent and ongoing trials have investigated a variety of combination chemotherapeutic regimens (variously employing ifosfamide, doxorubicin, gemcitabine, temozolomide, vincristine, cisplatin, and dacarbazine, among others) as well as targeted therapies, which in some cases have yielded improvements in response rate but which have had little impact on survival. No other medical option is currently available, and the median survival of patients with soft-tissue sarcoma with non-resectable metastases is around 12-15 months, and approximately 8 months after second line chemotherapy.

Liposarcomas are STS which account for at least 20% of all STS in adults. They can be further classified into 3 histologically and biologically different subtypes: well-differentiated liposarcoma/dedifferentiated liposarcoma (ALT-WD), myxoid or round cell liposarcoma and pleomorphic liposarcoma.

ALT-WD liposarcomas are locally aggressive rarely metastasizing tumors characterized by ring or giant marker chromosomes on the cytogenetic analysis and by amplification of the 12q13-21 region on Fluorescence In Situ Hybridization (FISH) (MDM2, CDK4 and HMGIC). They account for about 40% iv of liposarcomas with a 5 year Overall survival (OS) around 80%. In a series of WD/DD treated with several regimens response rate was 12.5% OS 15 months and median PFS 3.6 months(95 confidence interval (CI): 3.3-5.9) Mixoid /round cell liposarcoma accounts for 45-50% of all liposarcomas. They tend to metastasize to unusual soft tissue and bone locations. High histologic grade with more than 5% of round cell component is associated with a 5-year OS of 50% approximately. They are characterized by t(23;16)(q13-14;p11) which leads to the fusion of CHOP and TLS genes Pleomorphic liposarcoma accounts for approximately 5-10% of all liposarcomas, characterized by high grade features with frequent and early lung metastasis and cytogenetically by high chromosome counts and complex structural rearrangements.

VEGF is expressed in many STS in which increased expression is associated with higher grade and worse prognosis.

Pazopanib is an oral angiogenesis inhibitor that targets mainly VEGFR, PDGFR and c-kit. Recently the results of a phase II trial of pazopanib in STS have been published. It was a four-cohort 2-stages study. The liposarcoma stratum was closed after the first stage because of a PFS at 12 weeks of 17% (3 out of 17 patients did not progressed after 12 weeks). After central pathologic review, 2 other patients initially classified as other STS were found to have liposarcoma with stable disease at 12 weeks (5/19: 26% PFS12w), thus fulfilling criteria for cohort expansion. Phase II study had been completed and in phase III study patients with liposarcomas were excluded so therefore data on the liposarcoma cohort are inconclusive.

Furthermore the positive results of the phase III study PALETTE have been recently communicated, encouraging this treatment in other sarcomas: progression-free survival (PFS) per independent review was significantly prolonged with pazopanib (median: 4.6 vs 1.5 months; HR=0.31, 95% CI 0.24-0.40; P<0.0001). The interim analysis for overall survival shows a statistically non-significant improvement of pazopanib vs placebo (median: 11.9 vs 10.4 months, HR=0.83, 95% CI 0.62-1.09).

Soluble factors associated with efficacy and toxicity of pazopanib in these patients had been also reported. Decreases in VEGFR2 and increase in PlGF were both associated with toxicity (HTA and TSH elevation) and poorer prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up.

   Informed consent must be obtained prior to start of the specified screening window.

   Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study such as bone scan) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.
2. Age ≥ 18 years or legal age of consent if greater than 18 years
3. Histological confirmed diagnosis of high or intermediate grade malignant liposarcoma with metastatic or locally advanced disease. Formalin fixed paraffin embedded tumour block and/or representative H/E (haematoxylin/eosin) slides must be available for central pathologic review to classify tumors in the 2 eligible subtypes:

   Well-differentiated liposarcoma/de-differentiated liposarcoma (ALT-WD) Myxoid/round cell liposarcoma
4. Patient must have documentation of disease progression within 6 months prior to study entry.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Measurable disease by RECIST v1.1 criteria. At least one measurable lesion located outside of a previously irradiated area. If the only measurable lesion is in a previously irradiated area, RECIST progression should be documented after radiotherapy, in the previous 6 months before study entry.
7. The patient should not be considered eligible for surgery or radical radiotherapy. e.g. Patients to whom surgery/radiotherapy can not be performed with a curative intent due to the extension of the disease. In the case of radiotherapy, it may also be limited due to a previous treatment with radiotherapy in the same area.
8. The patient must have either been considered ineligible for systemic chemotherapy or received at least one previous regimen for relapsed, refractory or metastatic disease. A maximum of three previous lines for advanced/metastatic disease are allowed.

   Patients not eligible for systemic chemotherapy:

   Because of age, a biological condition or patient-refusal Generally, patients that received anthracyclines in the adjuvant setting are not eligible for first line therapy with this agent for advanced disease.

   Patients with a solitary kidney or >60 years old are usually not the best candidates for treatment with regular doses of ifosfamide.
9. Tumor tissue must be provided for all subjects for biomarker analysis before/during treatment with investigational product.
10. The patient should be able to swallow and retain study drug
11. Adequate organ system function as defined:

    Absolute neutrophil count (ANC)≥ 1.5 X 109/L Hemoglobin ≥ 9 g/dL (5.6 mmol/L) Platelets ≥ 100 X 109/L Prothrombin time (PT) or international normalized ratio (INR)≤ 1.2 X ULN Activated partial thromboplastin time (aPTT)≤ 1.2 X ULN Total bilirubin≤ 1.5 X ULN Alanine amino transferase (ALT) and Aspartate aminotransferase (AST) ≤ 2.5 X ULN Serum creatinine ≤ 1.5 mg/dL (133 µmol/L)Or, if >1.5 mg/dL: Calculated creatinine clearance (ClCR)≥ 30 mL/min to ≥ 50 mL/min Urine Protein to Creatinine Ratio (UPC) <1 Or, 24-hour urine protein <1g
    1. Subjects may not have had a transfusion within 7 days of screening assessment.
    2. Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.
    3. Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted.
    4. If UPC ≥ 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1 g to be eligible. Use of urine dipstick for baseline renal function assessment is not acceptable.
12. A female is eligible to enter and participate in this study if she is of:

    Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

    A hysterectomy A bilateral oophorectomy (ovariectomy) A bilateral tubal ligation Is post-menopausal Female subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L).

    Female subjects using HRT must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT

    Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. The acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

    Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product Oral contraceptive, either combined or progestogen alone Injectable progestogen Implants of levonorgestrel Estrogenic vaginal ring Percutaneous contraceptive patches Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository) Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug
13. LVEF above the lower limit of normal for the institution, based on ECHO or MUGA.

Exclusion Criteria:

1. Prior history of malignancies other than liposarcoma. Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
2. Clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
3. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   Active peptic ulcer disease Known intraluminal metastatic lesion/s with risk of bleeding Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
4. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

   Malabsorption syndrome Major resection of the stomach or small bowel.
5. Corrected QT interval (QTc) > 480 msecs
6. History of any one or more of the following cardiovascular conditions within the past 6 months:

   Cardiac angioplasty or stenting Myocardial infarction Unstable angina Coronary artery bypass graft surgery Symptomatic peripheral vascular disease Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
7. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].

   Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement. These three values should be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure. The mean SBP / DBP ratio must be <140/90 mmHg (OR 150/90 mm Hg, if this criterion is approved by Safety Review Team) in order for a subject to be eligible for the study.
8. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

   Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
9. Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
10. Evidence of active bleeding or bleeding diathesis.
11. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.

    Lesions infiltrating major pulmonary vessels (contiguous tumour and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessels is acceptable (CT with contrast is strongly recommended to evaluate such lesions).
12. Recent hemoptysis (≥ ½ teaspoon of red blood within 8 weeks before first dose of study drug).
13. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
14. Unable or unwilling to discontinue use of prohibited medications listed in section 7.4 of this protocol or at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
15. Treatment with any of the following anti-cancer therapies:

    radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of Pazopanib chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of Pazopanib
16. Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment
17. Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01-29 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Valverde, MD, Study Chair — Hospitals de la Vall de Hebron; Bernd Kasper, MD, Principal Investigator — University Medical Centre Mannheim
Locations (15):
- Germany (5):
  - HELIOS Klinikum Berlin-Buch (Sarkomzentrum Berlin-Brandenburg), Berlin
  - Universitätsklinikum EssenInnere Klinik (Tumorforschung), Essen
  - Medizinische Hochschule Hannover (Zentrum Innere Medizin), Hanover
  - Universitätsmedizin Mannheim (Sarkomzentrum), Manheim
  - Klinikum Großhadern der LMU Universität München (Med. Klinik und Poliklinik II), Munich
- Spain (10):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Canary Islands
  - Hospital de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2013 to 2018, advanced and/or metastatic liposarcoma patients were recruited across 12 centres from Spain and Germany.
Pre-assignment Details: Patients were clustered in two cohorts based on the liposarcoma type:
  * Cohort A: well differentiated liposarcoma
  * Cohort B: Myxoid/round cell liposarcoma
  Both cohorts were included in the single arm treatment: Pazopanib
Period: Overall Study
Arm/Group | Pazopanib
Started | 52
3 Weeks Pazopanib (Per Protocol PP) | 50
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 13
  Spain | 39
Height [Median (Standard Deviation); unit: cm] | 168.1 (11.1)
Body weight [Median (Standard Deviation); unit: Kg] | 77.3 (14.2)
Systolic pressure [Median (Standard Deviation); unit: mm Hg] | 132.5 (15.9)
Diastolic pressure [Median (Standard Deviation); unit: mm Hg] | 78.8 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Assessed 12 Weeks After Start of Treatment
Description: The primary objective of this study is to evaluate the activity of Pazopanib in patients with advanced and/or metastatic liposarcoma by means of progression-free survival (PFS) assessed 12 weeks after start of treatment. (According the RECIST criteria 1.1 and central radiology review).
  Progression was defined according to RECIST criteria 1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 12 weeks after start of treatment
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 50
percentage of participants
  Cohort A: number analyzed (Participants) | 37
  Cohort A | 54.1 [38 to 70.2]
  Cohort B: number analyzed (Participants) | 13
  Cohort B | 46.2 [19.1 to 73.3]

2. Secondary Outcome: Overall Progression Free Survival (Median PFS)
Description: Overall progression free survival will be computed from the date of start of treatment to the first documented date of progression or the date of death, whatever the cause. Patients alive and free from progression at the time of the analysis will be censored at the date of last follow-up.
Time Frame: Imaging studies repeated every 6 weeks for the first 12 weeks and every 8 weeks up to 36 months.
Population: Per protocol
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pazopanib
Number analyzed (Participants) | 50
Weeks
  Pazopanib | 12.14 [7.75 to 16.53]
  Cohort A: number analyzed (Participants) | 37
  Cohort A | 15 [8.19 to 21.8]
  Cohort B: number analyzed (Participants) | 13
  Cohort B | 10.29 [5.09 to 15.49]

3. Secondary Outcome: Percentage of Patients With Objective Tumor Response (OR)
Description: Objective tumor response, measured according to the RECIST 1.1 criteria (central reviewing) at 6 and 12 weeks.
  Response criteria are essentially based on a set of measurable lesions identified at baseline as target lesions, and followed until disease progression.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 6 weeks and 12 weeks
Population: Per protocol (PP)
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Pazopanib
Number analyzed (Participants) | 50
Percentage of patients
  6 weeks OR (PP population) | 8 [0.5 to 15.5]
  12 weeks OR (PP population) | 4 [1.4 to 9.4]

4. Secondary Outcome: Overall Survival (OS)
Description: It will be computed from the date of start of treatment to the date of death, whatever the cause. Patients alive or lost for follow-up at the time of the analysis will be censored at the date of last follow-up.
Time Frame: Every 12 weeks from disease progression up to 36 months.
Population: Per protocol
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pazopanib
Number analyzed (Participants) | 50
Weeks
  Pazopanib | 70.43 [44.92 to 95.94]
  Cohort A: number analyzed (Participants) | 37
  Cohort A | 70.43 [42.69 to 98.1]
  Cohort B: number analyzed (Participants) | 13
  Cohort B | 71.29 [31.21 to 111.36]

5. Secondary Outcome: Clinical Benefit Rate
Description: Patients who achieve complete response (CR), partial response (PR), or stable disease (SD) for 6 months or more and an improvement of symptoms will be considered as having derived clinical benefit.
Time Frame: Imaging studies required to investigate known disease should be repeated every 6 weeks for the first 12 weeks and every 8 weeks up to 36 months.
Population: Per population
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Pazopanib
Number analyzed (Participants) | 50
Percentage of patients
  Pazopanib | 26 [13.8 to 38.2]
  Cohort A: number analyzed (Participants) | 37
  Cohort A | 32.4 [17.3 to 47.5]
  Cohort B: number analyzed (Participants) | 13
  Cohort B | 7.7 [6.8 to 22.2]

6. Secondary Outcome: Growth Modulation Index (GMI)
Description: GMI is the ratio between time to progression (TTP) with pazopanib (TTPp) divided by the TTPp-1 with the previous line of therapy.
  GMI index values higher than 1 indicate that Pazopanib treatment has an increased time to progression when compared to previous line of treatment.
  GMI index values lower than 1 indicate that Pazopanib treatment has a reduced time to progression when compared to previous line of treatment.
  Higher GMI values are associated to a better outcome.
Time Frame: Imaging studies required to investigate known disease should be repeated every 6 weeks for the first 12 weeks and every 8 weeks up to 36 months. At patient progression confirmed by means RECIST criteria V 1.1
Population: Per protocol with TTP and TTPp registered
Measure: Median (95% Confidence Interval); unit: Arbitrary units
Arm/Group | Pazopanib
Number analyzed (Participants) | 37
Arbitrary units
  Pazopanib | 0.4 [0.1 to 18.6]
  Cohort A: number analyzed (Participants) | 27
  Cohort A | 0.7 [0.1 to 18.6]
  Cohort B: number analyzed (Participants) | 10
  Cohort B | 0.2 [0.1 to 1.1]

7. Secondary Outcome: Safety Profile (According CTCAE, Version 4.0)
Description: The safety and tolerability of Pazopanib will be determined by means of type, incidence, severity, timing, seriousness, and relatedness; of reported adverse events (AEs), physical examinations, and laboratory tests. Toxicity will be graded and tabulated by the NCI-CTCAE v 4.0.
Time Frame: Every week during the first month, week 6, week 9, week 12, every 4 weeks until end of treatment and at the end of treatment visit (28 days after the end of treatment), up to 36 months
Population: Intention to treat
Measure: Number; unit: Patients
Arm/Group | Pazopanib
Number analyzed (Participants) | 52
Patients
  AEs Pazopanib | 52
  AEs Cohort A: number analyzed (Participants) | 37
  AEs Cohort A | 37
  AEs Cohort B: number analyzed (Participants) | 15
  AEs Cohort B | 15
  related AEs Pazpanib | 46
  related AEs Cohort A: number analyzed (Participants) | 37
  related AEs Cohort A | 33
  related AEs Cohort B: number analyzed (Participants) | 15
  related AEs Cohort B | 13
  AE grade ≥3 Pazopanib | 26
  AE grade ≥3 Cohort A: number analyzed (Participants) | 37
  AE grade ≥3 Cohort A | 17
  AE grade ≥3 Cohort B: number analyzed (Participants) | 15
  AE grade ≥3 Cohort B | 9
  related-AE grade ≥3 Pazopanib | 16
  related-AE grade ≥3 Cohort A: number analyzed (Participants) | 37
  related-AE grade ≥3 Cohort A | 11
  related-AE grade ≥3 Cohort B: number analyzed (Participants) | 15
  related-AE grade ≥3 Cohort B | 5
  prior to treatment AE Pazopanib | 44
  prior to treatment AE Cohort A: number analyzed (Participants) | 37
  prior to treatment AE Cohort A | 31
  prior to treatment AE Cohort B: number analyzed (Participants) | 15
  prior to treatment AE Cohort B | 13

ADVERSE EVENTS:
Time Frame: AEs up to 30 days after administration of the last dose of study drug, approximately 36 months
Description: Additionally to AEs and SAEs definitions, an abnormal objective test finding should be reported as an AE as follows:
  * test result associated with clinically significant symptoms
  * test result lead to a change in study dosing or discontinuation from the study, significant additional concomitant drug treatment or other therapy
  * test result leads to any of the outcomes included in the definition of a SAE
  * test result were considered to be an AE by the investigator
Arm/Group | Pazopanib
All-Cause Mortality (participants affected / at risk) | 35/52
Serious Adverse Events (participants affected / at risk) | 14/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib (N=52)
Abscess of tumor mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ALT increased (Blood and lymphatic system disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Ascites (General disorders) | 1 (1)
General status deterioration (General disorders) | 1 (1) — Fatal
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) — Fatal
Cardiac dysrhythmia (Cardiac disorders) | 1 (1)
Febrile neutropenia (Immune system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Femure fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac disorders (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Bilirrubin increase (Blood and lymphatic system disorders) | 1 (1)
Uncontrolled pain (General disorders) | 1 (1)
Tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor debulking (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=52)
Adverse Events (General disorders) | 52 — 52 patients presented adverse events, the list of adverse events by type was not further analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-02-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT01692496/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT01692496/SAP_001.pdf